CLINICAL TRIAL: NCT03643653
Title: The Establishment of China Bronchiectasis Registry and the Optimal Treatment Research Collaboration for Bronchiectasis (BEChina)
Brief Title: The Establishment of China Bronchiectasis Registry and Research Collaboration
Acronym: BEChina
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Collaborators: Ruijin Hospital (Other); Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Jin-Fu Xu, Chief of Respiratory and Critical Care Medicine, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: 20180814
Record Dates: First submitted 2018-08-16; First posted 2018-08-23 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; multi-centered registry
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Whole blood would be drawn and stored at - 80℃
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators meant to establish a multi-centered bronchiectasis patient registry for Chinese bronchiectasis patients. This would be the first bronchiectasis registry in China. Patients with all kinds of bronchiectasis would be enrolled.

DETAILED DESCRIPTION:
A multi-centered bronchiectasis patient registry would be founded, which will include patients from three teaching hospital (Ruijin Hospital, Zhongshan Hospital and Shanghai Pulmonary Hospital) in Shanghai at the beginning. The network will be promoted to other cities and different places in China. Patients with bronchiectasis would be enrolled and detailed information would be recorded. Follow-up of patients would provide more information on the prognosis of disease. Optimal treatment studies for the patients will be initiated one by one based on the network. The investigators are committed to promoting clinical research and education in bronchiectasis, through sharing of protocols, research idea and expertise.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with bronchiectasis according to 'non-cystic fibrosis bronchiectasis guideline' published by British Thoracic Society in 2010.
* Patients who are willing to sign the consent form and participate in the study.

Exclusion Criteria:

* Patients with incomplete essential information, which is needed for the integrity of data analysis. Essential information include CT images, respiratory sample cultures, spirometry and exacerbation history for at least one year.
* Patients under 18 years old.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with all-cause bronchiectasis would be included, such as those with tuberculosis history and genetic disorders.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients enrolled in the registry | 3 years
  To establish a multi-centered bronchiectasis registry in Shanghai

SECONDARY OUTCOMES:
Lung Function (FEV1, FVC, FEV1% pred, FVC% pred etc.) | recorded at baseline and re-tested every year, up to 3 years.
  Lung function would be tested by spirometry when patients visit the clinic.
Exacerbation | up to 3 years
  Exacerbation was defined as the use of antibiotics or even hospitalization due to the worsening of symptoms or emergence of new symptoms.
Aetiology | at baseline
  To analysis the possible cause of bronchiectasis in Shanghai, China.
Microbiology | At least 1 year before enrollment and 3 years during the follow-up
  Sputum or bronchoalveolar lavage fluid culture
Comorbidity | At baseline and updated every year for up to 3 years
  Comorbidity would be recorded.
Quality of Life Questionnaire-Bronchiectasis | At baseline and updated once a year for 3 years
  The questionnaire asks patients questions about their current state of health. It could be downloaded from the website online.
Bronchiectasis severity Score (BSI) | At baseline and updated once a year for 3 years
  The scale is presented online. It consists of 9 items including Age, BMI(Body Mass Index), % FEV1 Predicted, Previous Hospital Admission in the past 2 years, number of exacerbations in previous year, MRC Breathlessness Score, Pseudomonas Colonisation, Colonisation with other organisms,affected lobes.
  0-4 Mild Bronchiectasis. 5 - 8 Moderate Bronchiectasis. 9 + Severe Bronchiectasis.
E-FACED score | At baseline and updated once a year for 3 years
  It consists of 6 items including exacerbation history in the past year, % FEV1 predicted, Age, Chronic colonization by Pseudomonas aeruginosa, n° of pulmonary lobes affected,and Dyspnea (measured by mMRC score) mild: 0-3 points, moderate: 4-6 points; and severe: 7-9 points
Mortality | 3 years
modified Medical Research Council (mMRC) dyspnea score | At baseline and updated once a year for 3 years
  1. - Not troubled by breathlessness except on strenuous exercise
  2. - Short of breath when hurrying or walking up a slight hill
  3. - Walks slower than contemporaries on level ground because of breathlessness, or has to stop for breath when walking at own pace
  4. - Stops due to breathlessness after walking 100m
  5. - House bound due to breathlessness, or breathless on dressing or undressing.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Fu Xu, MD, Study Chair — Shanghai Pulmonary Hospital, Shanghai, China
Locations (2):
- China (2):
  - Shanghai Pulmonary Hospital , Tongji University, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chalmers JD, Aliberti S, Polverino E, Vendrell M, Crichton M, Loebinger M, Dimakou K, Clifton I, van der Eerden M, Rohde G, Murris-Espin M, Masefield S, Gerada E, Shteinberg M, Ringshausen F, Haworth C, Boersma W, Rademacher J, Hill AT, Aksamit T, O'Donnell A, Morgan L, Milenkovic B, Tramma L, Neves J, Menendez R, Paggiaro P, Botnaru V, Skrgat S, Wilson R, Goeminne P, De Soyza A, Welte T, Torres A, Elborn JS, Blasi F. The EMBARC European Bronchiectasis Registry: protocol for an international observational study. ERJ Open Res. 2016 Jan 20;2(1):00081-2015. doi: 10.1183/23120541.00081-2015. eCollection 2016 Jan. PMID 27730179
- [Derived] Gao YH, Lu HW, Mao B, Guan WJ, Song YL, Li YY, Wang DX, Wang B, Gu HY, Li W, Luo H, Wang LW, Li F, Guo FX, Zhang M, Jie ZJ, Hang JQ, Yang C, Ren T, Yuan Z, Meng QW, Jia Q, Chen Y, Chen RC, Qu JM, Xu JF. The Establishment of China Bronchiectasis Registry and Research Collaboration (BE-China): Protocol of a prospective multicenter observational study. Respir Res. 2022 Dec 3;23(1):328. doi: 10.1186/s12931-022-02254-9. PMID 36463140